CLINICAL TRIAL: NCT02192996
Title: Probiotic Supplementation to Improve the GUT Microbiota of Very Low Birth Weight, a Pilot Study
Brief Title: Probiotic Supplementation to Improve the GUT Microbiota of Very Low Birth Weight Preterm, a Pilot Study
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Hospital Universitario La Paz (Other)
Collaborators: Universidad Complutense de Madrid (Other)
Responsible Party: Principal Investigator, Esperanza Escribano, Medical doctor, Hospital Universitario La Paz
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: HULP3551; Universidad Complutense Madrid (Other: Academic)
Record Dates: First submitted 2014-06-24; First posted 2014-07-17 (Estimated); Last update posted 2014-07-17 (Estimated); Status verified 2014-07

CONDITIONS: Other Preterm Infants; NEC
Keywords: VLBW preterm; GUT microbiota; probiotics supplementation; immune compounds
MeSH Terms: interventions — Probiotics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Probiotics supplementation (Other): Five very low birth weight (VLBW) infants enrolled within 2 days of birth, with a weight < 1300 g and gestational age < 29 weeks and without any malformation or metabolic disease at birth were supplemented with two daily doses of a mixture of "Bifidobacterium breve" and "Lactobacillus salivarius" , probiotic strains isolated from human milk during their first weeks of life. The lyophilized powder has contained at least 1x10^9 colony forming units (CFU) per doses of each one of the probiotic bacteria.
  Interventions: Dietary Supplement: Probiotic

INTERVENTIONS:
Dietary Supplement: Probiotic — blood and fecal samples were collected from five VLBW preterms which were supplemented with a probiotic mixture of Bifidobacterium breve / Lactobacillus salivarius isolated from human milk
  Other Names: "Bifidobacterium breve / Lactobacillus salivarius mixture"

SUMMARY:
This pilot trial is designed to investigate the benefits of the use of probiotics in GUT microbiota development and/or immunological biomarkers and how this can be related with the clinical status of very low birth weight preterms during their first weeks of life at the neonatal intensive care unit(NICU).

DETAILED DESCRIPTION:
This pilot trial is designed to investigate the benefits of the use of mixtures of probiotics isolated from human milk in GUT microbiota development and/or immunological biomarkers. Furthermore, the relationship between evaluated parameters and the clinical status of very low birth weight preterms during their first weeks of life at the NICU will be analysed.

ELIGIBILITY:
Inclusion Criteria:

* preterm infants with birth weight less than one thousand and three hundred grammes
* preterm infants with gestational age less than 29 weeks

Exclusion Criteria:

* mayor malformations
* chromosomopathies
* congenital infections
* non parental consent

Ages: 1 Hour to 1 Week | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 5 (Actual)
Dates: Start 2012-12; Primary Completion 2013-02 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
changes in microbiological counts in feces of preterm infants | prior to initiate and at 7th, 14th, 21th, 28th days receiving probiotics
  Adequate dilutions of meconium and stool samples were spread onto general and selective culture media for the enumeration of different bacterial species. Identification of isolates was carried out by matrix-assisted laser desorption ionization-time of flight (MALDI-TOF) mass spectrometry.

SECONDARY OUTCOMES:
concentration of immunological parameters on feces | prior to star and at 7th, 14th and 21st days of receiving probiotics
  multiplex methodology and enzyme-Linked ImmunoSorbent Assay (ELISA) were used to determine a wide range of immune compounds and calprotectin as immune system status biomarkers: immunoglobulin(Ig) G1, IgG2, IgG3, IgG4, IgM, IgA, interleukin (IL)-1b, IL-6, IL-12,interferon-gamma, Tumor necrosis factor-alpha,IL-2,IL-4,IL-10, IL-13, IL-17, IL-8, growth related oncogene- alpha, macrophages chemoattractant protein-1, macrophage inflammatory protein-1b, IL-5, IL-7, granulocytemacrophage -colony stimulating factor (GM-CSF), granulocyte-colony stimulating factor (G-CSF).
concentration of immunological parameters on plasma samples | 7th, 14th, 19th and 24th days of receiving probiotic).
  multiplex methodology and enzyme-Linked ImmunoSorbent Assay (ELISA) were used to determine a wide range of immune compounds and calprotectin as immune system status biomarkers: immunoglobulin(Ig) G1, IgG2, IgG3, IgG4, IgM, IgA, interleukin (IL)-1b, IL-6, IL-12,interferon-gamma, Tumor necrosis factor-alpha,IL-2,IL-4,IL-10, IL-13, IL-17, IL-8, growth related oncogene- alpha, macrophages chemoattractant protein-1, macrophage inflammatory protein-1b, IL-5, IL-7, granulocytemacrophage -colony stimulating factor (GM-CSF), granulocyte-colony stimulating factor (G-CSF).

OTHER OUTCOMES:
clinical features during NICU stay | during NICU stay, arround 1 moth
  medical staff registered all the clinical status of the enrolled infants, after that the most relevant morbidity parameters associated to prematurity were factorized and evaluated by the clinicians, prior to evaluate the possible relationships with the other outcomes measured.
  -Necrotizing enterocolitis, late onset sepsis, intestinal motility evaluated by feeding tolerance and determination ot total gastrointestinal transit time by the administration of carmin red, type of feeding, respiratory support, intraventricular hemorrhage. Describe healthy status of each preterm

CONTACTS AND LOCATIONS:
Overall Officials: Miguel Saenz de Pipaon, PhD. MD., Principal Investigator — Hospital Universitario La Paz
Locations (1):
- Hospital Universitario La Paz, Madrid, Madrid, Spain